CLINICAL TRIAL: NCT03016832
Title: A Randomized, Double-blind, Parallel-controlled, Multi-center Clinical Trial of HuangKui Capsule to Treat Diabetic Kidney Disease
Brief Title: Clinical Trial of HuangKui Capsule to Treat Diabetic Kidney Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SZCT-2016-01
Record Dates: First submitted 2017-01-04; First posted 2017-01-11 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2016-12

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Irbesartan; Huangkui

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Huangkui (Experimental): Placebo drug that simulates Irbesartan tablets 150mg /qd, oral dosing; HuangKui Capsule 2.5g/tid, oral dosing
  Interventions: Drug: Placebo drug that simulates Irbesartan tablets; Drug: HuangKui Capsule
- controlled (Active Comparator): Placebo drug that simulates Irbesartan tablets 150mg /qd, oral dosing; HuangKui Capsule 2.5g/tid, oral dosing irbesartan tablets 150mg /qd, oral dosing; Placebo drug that simulates HuangKui capsule 2.5g/tid, oral dosing
  Interventions: Drug: irbesartan tablets; Drug: Placebo drug that simulates HuangKui capsule
- combined treatment (Other): irbesartan tablets 150mg /qd, oral dosing HuangKui Capsule 2.5g/tid, oral dosing.
  Interventions: Drug: irbesartan tablets; Drug: HuangKui Capsule

INTERVENTIONS:
Drug: Placebo drug that simulates Irbesartan tablets — Placebo drug that simulates Irbesartan tablets 150mg /qd, oral dosing
  Arms: Huangkui
Drug: irbesartan tablets — irbesartan tablets 150mg /qd, oral dosing
  Arms: combined treatment; controlled
Drug: Placebo drug that simulates HuangKui capsule — Placebo drug that simulates HuangKui capsule 2.5g/tid, oral dosing
  Arms: controlled
Drug: HuangKui Capsule — HuangKui Capsule 2.5g/tid, oral dosing.
  Arms: Huangkui; combined treatment

SUMMARY:
1. Name of Investigational Products Huangkui capsule.
2. Trial Topic A Randomized, Double-blinded, Parallel, controlled, Multicenter Clinical Trial of Huangkui Capsule in Treating Type II Diabetic Nephropathy (DKD)
3. Trial Objectives Primary objective:To evaluate HuangKui capsule efficacy for treatment of type II diabetes ACR.

   Secondary objective: To evaluate the efficacy of HuangKui capsule on 24-hour urinary protein changes、reduce PCR-increase eGFR, improve micro-inflammatory state, and improving Traditional Chinese medicine clinical efficacy
4. Trial Design Designed as a block randomized, double-blinded, parallel controlled, multi-center clinical trial.

DETAILED DESCRIPTION:
1. Name of Investigational Products Huangkui capsule
2. Trial Topic A Randomized, Double-blinded, Parallel, controlled, Multicenter Clinical Trial ofHuangkui Capsule in Treating Type II Diabetic Nephropathy (DKD)
3. Trial Objectives Primary objective: To evaluate HuangKui capsule efficacy for treatment of type II diabetes ACR.

   Secondary objective: To evaluate the efficacy of HuangKui capsule on 24-hour urinary protein changes、reduce PCR-increase eGFR, improve micro-inflammatory state, and improving Traditional Chinese medicine clinical efficacy.
4. Trial Design Designed as a block randomized, double-blinded, parallel controlled, multi-center clinical tria 4.1 Multi-center: The trial is proposed to be conducted in the department of Nephrology or Endocrinology of nine hospitals simultaneously.

   4.2 Randomization:Using stratified block randomized design. The randomization numbers were generated with SAS statistical software.

   4.3 Arms: The study subjects were divided into 3 arms: Huangkui arm, controlled arm and combined treatment arm.

   4.4 Estimation of subject numbers

   This study was based on the main indicator ACR to calculate the sample size, according to the clinical protocol:

   ①The change of ACR of Irbesartan combined with Huangkui capsule is superior than Irbesartan monotherapy.

   ②The changes of ACR in the monotherapy group were significantly lower than those in the irbesartan monotherapy group According to the experience of clinical treatment, it was found that the change of ACR was about 12.85mg / g before treatment with Irbesartan combined with Huangkui capsule group and 6.50mg / g before and after treatment with Irbesartan group, and α = 0.05 (bilateral (1-β) = 80%, the standard deviation of the change value before and after ACR treatment with irbesartan combined with Huangkui capsule group was 17.18, Check the sample size calculation formula The number of samples in each group was calculated as n western medicine group = n combined treatment group = 110 cases.

   Another group based on the clinical treatment experience to take the standard deviation of 17.18, take α = 0.025 (unilateral test), β = 0.2, that is, the degree of control (1-β) = 80% of the case, the non-inferior boundary value of 6.50mg / g, according to the non-inferior test sample size calculation formula, The number of samples in each group was calculated as n western medicine group = n Chinese traditional treatment group = 110 cases.According to the program requirements, the three groups were designed to be 1: 1: 1, taking into account the blanding method and 20% rejection rate. ultimately a total of 414 cases included in the case, each group of 138 cases.

   4.5 Blinding: double-blinding. Blinding will be conducted by statisticians as two levels of blinding. Level 1 Blinding: blinding of the investigational products. The investigational products and comparative products use unified packaging; level 2 blinding: the blinding of the packaging box of investigational products.
5. Diagnostic criteria The etiology of Diabetic nephropathy is kidney damage, referred to DN in the past (diabetic nephropathy). But in 2007, the American Foundation for Kidney Disease (NKF) developed guidelines for the life quality of kidney disease (NKF / KDOQI). The guidelines recommend that DKD (diabetic kidney disease) instead of DN. In 2014, the American Diabetes Association (ADA) and NKF reached a consensus that DKD referred to the chronic kidney disease caused by diabetes, including glomerular filtration rate (GFR) which is less than 60ml.min-1.1.73m-2 or urine white Protein / creatinine ratio (ACR) is higher than 30 mg / g for more than 3 months,associated with diabetic retinopathy.

   During having diagnosis, if one of the following circumstances happened, we should consider its CKD is caused by (1) no diabetic retinopathy; (2) GFR lower or decreased rapidly; (3) a sharp increase in proteinuria or nephrotic syndrome; (4) refractory hypertension; (5) urinary sediment activity;(6) symptoms or signs of other systemic diseases; (7) glomerular filtration rate decreased by more than 30% within 2-3 months after initiation of treatment with angiotensin converting enzyme inhibitors (ACEI) or angiotensin II receptor antagonists (ARB).

   5.2 Table of TCM symptom/signs Diagnostic dosage It is refer to "Clinical research guidelines of new drug of Traditional Chinese Medicine "(2002 version), which published by China Medical Science andTechnology Press
6. Treatment options 6.1 Basic treatment 6.1.1 Anti-hypotensive We can choose antihypertensive drugs Monotherapy or combined controling blood pressure expect ACEI and ARB, control blood pressure in 160 / 90mmHg the following 6.1.2 Anti-hypoglycemic We can use oral hypoglycemic agents or insulin for hypoglycemic, so that glycosylated hemoglobin ≤ 8.5%.

   6.1.3 Anti-hypolipidemic We can choose to use statins or fibrates lipid-lowering drugs. 6.1.4 Diet control Patients with edema should limit the salt and water, daily sodium intake <5g; high protein diet increased glomerular hyperperfusion, high filtration, and therefore advocated the principle of high quality low-protein diet. Protein intake should be a high biological value of animal protein-based, early protein intake should be limited to 1g/（kg•d） 6.2 Investigational products Huangkui Capsule: produced by SZYY Group Pharmaceutical Limited, Jiangsu, 0.5g×30 capsules/box Placebo that simulates Huangkui capsule: produced by SZYY Group Pharmaceutical Limited, 0.5g×30 capsules/box Irbesartan tablets: produced by Sanofi (Hangzhou) Pharmaceutical Co., Ltd., 150mg×7 capsules/box Placebo that simulates Irbesartan tablets: produced by SZYY Group Pharmaceutical Limited, Jiangsu, 150mg×7 capsules/box 6.3 Trial process 6.3.1 Treatment for observation period The subjects who meet the inclusion criteria will be randomized into three groups at a 1:1:1 ratio.

   Test group: Placebo drug that simulates Irbesartan tablets 150mg /qd, oral dose; Huangkui Capsule 2.5g/tid, oral dose.

   Control group: irbesartan tablets 150mg /qd, oral dose; Placebo drug that simulates Huangkui capsule 2.5g/tid, oral dose.

   Combined treatment group: irbesartan tablets 150mg /qd, oral dose; Huangkui Capsule 2.5g/tid, oral dose.

   6.3.2 period of treatment Treatment observation period is 24 weeks, follow-up points: Week 0, 4, 8, 12, 16, 20, 24.

   6.4 Concomitant medications During the import period and throughout the treatment, do not use the RAS blockers (ARB or ACEI) other than the investigational product irbesartan and Potassium-sparing diuretics, Calcium dobesilate, Aldehyde-containing starch, or other Chinese medicine which can reduce proteinuria.

   If other medicines have been used before the trial, the subjects can continue to use them. The use of these medicines should be recorded.

   6.5 ACR Detection Specimens: one - time morning urine (after 5:00); Urinary creatinine detection method: enzyme kinetics; urinary albumin detection method : immune turbidimetric method. 6.6 PCR detection Specimens: 24h urine Urine creatinine detection method: Enzyme kinetic method Urine protein detection method: dye binding method PCR = urinary protein / creatinine
7. Efficacy endpoint 7.1 Efficacy endpoint 7.1.1 Primary endpoints ACR baseline changes and changes in the rate 7.1.2 Secondary endpoints （1）24-hour urinary protein quantification baseline changes and changes in the rate （2）PCR baseline changes and changing rate （3）Glomerular filtration rate (eGFR)baseline changes （4）High sensitivity C - reactive protein baseline values （5）TCM syndromes Efficacy endpoint Changes and the rate change before and after treatment. [Time point: baseline,12-weeks treatment,24-weeks treatment]

   7.2 Efficacy endpoint Evaluation endpoints 7.2.1 The ACR change rate ( refer to "Guiding principles of clinical research on the treatment of chronic nephritis with traditional Chinese medicine", 2002 version; The State Administration of Traditional Chinese Medicine in 1987 to develop the Efficacy endpoint of chronic glomerulonephritis standard ) Complete remission: ACR is less than 30mg/g; Markedly effective: ACR decreased more than 50% before treatment Effective: ACR decreased more than 30%-50% before treatment Invalid: those who did not meet these targets. 7.2.2 Efficacy endpoint for TCM syndrome Changes in value and rate before and after treatment before and after treatment [Time point: baseline,12-weeks treatment,24-weeks treatment]
8. Safety Evaluation endpoints 8.1 Vital signs, such as such as body temperature, pulse, breathing, blood pressure and so on.

   8.2 Blood, urine routine test, liver function test(ALB、ALT、AST), renal function test(Bun、SCr, UA、eGFR), electrocardiogram, blood potassium, blood sugar; Adverse events/adverse reactions.
9. Statistical Methods All statistical calculations were carried out using SAS v9.3 statistical analysis software, hypothesis testing are used bilateral test, unless otherwise specified, the overall comparison between the test level = 0.05.

Statistical analysis includes：Three groups of subjects enrolled No., drop out and excluded cases, demographic and other baseline characteristics, compliance, efficacy analysis and safety analysis.

For quantitative data, we conduct descriptive statistical analysis with cases, averages, standard deviation, minimum, median, maximum, upper quartile (Q1), lower quartile (Q3) and 95% confidence interval (95% CI). Comparisons between treatment groups were performed using either an analysis of variance or a Wilcoxon rank sum test. If the influence of covariates is taken into account, a general linear model (GLM) is used.

Descriptive statistical analysis of qualitative data is given in terms of the number of cases and their percentages. Count data were compared between each treatment group, using x2 test, Fisher exact probability method; grade data in each treatment group or between groups before and after treatment comparison analysis, Wilcoxon rank sum test. If the effects of the center or other factors are taken into account, a CMH x2 test or Logistic regression is used.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years old, male or female
2. Meet the diagnostic criteria of type 2 diabetes published by the World Health Organization (WHO) in 1999: fasting plasma glucose>126mg/dL (or>7.0mmol/L), 2h postprandial blood glucose>200mg/dL (or>11.1mmol/L), or 2h blood glucose in OGTT test>200mg/dL(11.1mmol/L), random blood glucose test≥200mg/dL(11.1mmol/L)
3. Meet Diabetic Kidney Disease (DKD) and the United States Diabetes Association (ADA) and the American Kidney Foundation (NKF) diagnostic criteria in 2007 ; 300mg/g ≤ ACR <2000mg/g
4. e-GFR>30 mL/min (CKD-Epi formula),
5. Glycated hemoglobin ≤8.5%
6. Agree to sign informed consent form.

Exclusion Criteria:

1. Type 1 diabetes
2. Other secondary glomerulonephritis caused by Non-diabetes disease;
3. Taking Huangkui capsule, ACEI and / or ARB drugs within 2 months;
4. Taking glucocorticoid, immunosuppressive agents and Tripterygium wilfordii drug history within one month;
5. Taking three or more antihypertensive drugs, but the blood pressure is still>160/90mmHg
6. With other diseases, syndromes, or comorbidities that may affect the diagnosis and therapeutic effect of the target indications
7. The treatments received may affect the evaluation of efficacy and safety endpoints
8. With phychological or pathological conditions which may affect the evaluation of efficacy endpoints and safety endpointssuch as the menstrual period, or heart, brain, liver and hematopoietic system and other serious primary disease
9. With high risk, such as pregnant women or childbearing during the trial, be allergy to the Abelmoschus Moschatus Capsule and irbesartan, in the dangerous condition with unexpected accidents.
10. Alcohol or drug abuse
11. Noncompliance, such as unwilling to accept research procedures or suffering from mental illness and other diseases
12. Other: Such as poor compliance, or can not attend the follow-up visit in time for some reasons;
13. Is participating in another clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-05 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
ACR | every 4 week，a total of 24 weeks
  ACR baseline changes and changes in the rate

SECONDARY OUTCOMES:
24-hour urinary protein | every 4 week,，a total of 24 weeks
  24-hour urinary protein quantification baseline changes and changes in the rate
PCR | every 12 week,，a total of 24 weeks
  PCR baseline changes and changing rat
Glomerular filtration rate | every 12 week,，a total of 24 weeks
  Glomerular filtration rate (eGFR) baseline changes
TCM syndromes Efficacy endpoint | baseline,12-weeks treatment,24-weeks treatment
  Changes and the rate change before and after treatment.
High sensitivity C | baseline,12-weeks treatment,24-weeks treatment
  High sensitivity C - reactive protein baseline values

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital of TCM, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhao J, Tostivint I, Xu L, Huang J, Gambotti L, Boffa JJ, Yang M, Wang L, Sun Z, Chen X, Liou-Schischmanoff A, Baumelou A, Ma T, Lu G, Li L, Chen D, Pieroni L, Liu B, Qin X, He W, Wang Y, Gu HF, Sun W. Efficacy of Combined Abelmoschus manihot and Irbesartan for Reduction of Albuminuria in Patients With Type 2 Diabetes and Diabetic Kidney Disease: A Multicenter Randomized Double-Blind Parallel Controlled Clinical Trial. Diabetes Care. 2022 Jul 7;45(7):e113-e115. doi: 10.2337/dc22-0607. No abstract available. PMID 35613364